CLINICAL TRIAL: NCT07302126
Title: Preventive Efficacy of Bergmann Enema for Acute Radiation-induced Rectal Injury in Rectal Cancer Patients Undergoing Short-course Radiotherapy: a Prospective, Single-arm, Phase II Trial
Brief Title: Preventive Efficacy of Bergmann Enema for Acute Radiation-induced Rectal Injury in Rectal Cancer Patients Undergoing Short-course Radiotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Berg-ARRI-SCRT
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Radiation Enteritis
Keywords: Acute radiation-induced rectal injury; Rectal cancer; Short-course radiotherapy; Bergmann enema
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention: Patients will receive Bergmann enema (30 ml) once daily from the start of radiotherapy until the 10th day after the end of radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients will receive Bergmann enema (30 ml) once daily from the start of radiotherapy until the 10th day after the end of radiotherapy.
  Interventions: Drug: Bergmann enema

INTERVENTIONS:
Drug: Bergmann enema — Patients will receive Bergmann enema (30 ml) once daily from the start of radiotherapy until the 10th day after the end of radiotherapy.

SUMMARY:
Research Objective and Principle: To evaluate the effectiveness of Bergmann enema in preventing acute radiation-induced rectal injury in patients with rectal cancer, thereby providing a basis for treatment options for potential radiation-induced rectal injury patients, aiming for adoption by international guidelines.

Primary Objective: Incidence of grade 2 or higher radiation-induced rectal injury.

Secondary Objectives: Severity of radiation-induced rectal injury, completion rate of short-course radiotherapy, safety of Bergmann enema, quality of life, pathological complete response (pCR) rate.

Study Design: Prospective, single-center, single-arm study.

Study Population and Expected Enrollment: Patients with rectal cancer undergoing short-course radiotherapy, expecting to enroll 40 patients.

Trial Duration: From December 2025 to December 2026.

Intervention: Patients will receive Bergmann enema (30 ml) once daily from the start of radiotherapy until the 10th day after the end of radiotherapy.

Statistical Hypothesis: Based on previous reports, the incidence of acute radiation-induced rectal injury is 80%, and it is expected that Bergmann enema preventive treatment can reduce it to 50%. The sample size was estimated using a formula designed to calculate single-group rate, with a set at 0.05 and a power of 80%. The study aimed to enroll at least 36 patients. Considering a dropout rate of 10%, at least 40 patients need to be included.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, regardless of gender;
2. Fully understand this study and voluntarily sign the informed consent form, able to comply with the study protocol and complete all trial procedures;
3. Patients with pathologically confirmed mid-lower rectal cancer;
4. Undergoing short-course pelvic radiotherapy (total dose of 25-35Gy in 5.0-7.0 fractions over 5 consecutinve days);
5. Eastern Cooperative Oncology Group (ECOG) score of 0-1, with an expected survival time of more than 6 months;
6. Assessment by the attending physician and researcher indicates that vital organ function can tolerate the treatment risks.

Exclusion Criteria:

1. Severe comorbidities, including uncontrolled stable medical diseases after treatment, or a history of neurological or psychiatric disorders (such as dementia or epilepsy), making them unsuitable for radiotherapy;
2. Patients who have received pelvic radiotherapy;
3. Presence of malignant pleural effusion or malignant abdominal effusion, or accompanied by bowel obstruction;
4. Pregnant or breastfeeding women;
5. Patients expected to undergo major surgery during the study period;
6. Participation in other clinical trials within 4 weeks prior to enrollment;
7. A history of alcohol abuse, drug use, or substance abuse within the past year;
8. Severe allergic constitution, or allergy to Bergmann;
9. Inability to cooperate with the enema;
10. Subjects deemed unsuitable for participation in this trial for other reasons by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher radiation-induced rectal injury | 3 months

SECONDARY OUTCOMES:
Severity of radiation-induced rectal injury | 3 months
Completion rate of short-course radiotherapy | 9 months
Safety of Bergmann enema | 9 months
Pathological complete response (pCR) rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennedy M, Bruninga K, Mutlu EA, Losurdo J, Choudhary S, Keshavarzian A. Successful and sustained treatment of chronic radiation proctitis with antioxidant vitamins E and C. Am J Gastroenterol. 2001 Apr;96(4):1080-4. doi: 10.1111/j.1572-0241.2001.03742.x. PMID 11316150
- [Result] Ehrenpreis ED, Jani A, Levitsky J, Ahn J, Hong J. A prospective, randomized, double-blind, placebo-controlled trial of retinol palmitate (vitamin A) for symptomatic chronic radiation proctopathy. Dis Colon Rectum. 2005 Jan;48(1):1-8. doi: 10.1007/s10350-004-0821-7. PMID 15690650
- [Result] 王楠, 丁田贵与尹立杰, 医用射线防护喷剂防治放射性口腔黏膜炎的临床观察. 口腔医学, 2020. 40(08): 第728-730+737页.
- [Result] 李祎萍, 医用射线防护喷剂应用在乳腺癌患者急性放射性皮肤损伤中的效果. 实用临床护理学电子杂志, 2016. 1(12): 第167+169页.
- [Result] 张力元等, 医用射线防护喷剂防治皮肤黏膜放射性损伤的临床观察. 中华放射医学与防护杂志, 2006(06): 第597-599页.
- [Result] 张慧, 章真与袁双虎, 放射性直肠损伤的预防与治疗临床实践指南. 中华肿瘤防治杂志, 2023. 30(5): 第245-259页.
- [Result] 中华医学会外科学分会结直肠外科学组, 中国医师协会外科医师分会结直肠外科医师委员会与中国抗癌协会大肠癌专业委员会, 中国放射性直肠损伤多学科诊治专家共识（2021版）. 中华胃肠外科杂志, 2021. 24(11): 第937-949页.
- [Result] 中国医师协会外科医师分会与中华医学会外科学分会结直肠外科学组, 中国放射性直肠炎诊治专家共识(2018版). 中华胃肠外科杂志, 2018. 21(12): 第1321-1336页.
- [Result] Paquette IM, Vogel JD, Abbas MA, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of The American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Treatment of Chronic Radiation Proctitis. Dis Colon Rectum. 2018 Oct;61(10):1135-1140. doi: 10.1097/DCR.0000000000001209. No abstract available. PMID 30192320
- [Result] Jahraus CD, Bettenhausen D, Malik U, Sellitti M, St Clair WH. Prevention of acute radiation-induced proctosigmoiditis by balsalazide: a randomized, double-blind, placebo controlled trial in prostate cancer patients. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1483-7. doi: 10.1016/j.ijrobp.2005.04.032. Epub 2005 Aug 15. PMID 16099600
- [Result] Gami B, Harrington K, Blake P, Dearnaley D, Tait D, Davies J, Norman AR, Andreyev HJ. How patients manage gastrointestinal symptoms after pelvic radiotherapy. Aliment Pharmacol Ther. 2003 Nov 15;18(10):987-94. doi: 10.1046/j.1365-2036.2003.01760.x. PMID 14616164
- [Result] Qin Q, Huang B, Cao W, Zhou J, Ma T, Zhou Z, Wang J, Wang L. Bowel Dysfunction After Low Anterior Resection With Neoadjuvant Chemoradiotherapy or Chemotherapy Alone for Rectal Cancer: A Cross-Sectional Study from China. Dis Colon Rectum. 2017 Jul;60(7):697-705. doi: 10.1097/DCR.0000000000000801. PMID 28594719
- [Result] Qin Q, Ma T, Deng Y, Zheng J, Zhou Z, Wang H, Wang L, Wang J. Impact of Preoperative Radiotherapy on Anastomotic Leakage and Stenosis After Rectal Cancer Resection: Post Hoc Analysis of a Randomized Controlled Trial. Dis Colon Rectum. 2016 Oct;59(10):934-42. doi: 10.1097/DCR.0000000000000665. PMID 27602924
- [Result] Haddock MG, Sloan JA, Bollinger JW, Soori G, Steen PD, Martenson JA; North Central Cancer Treatment Group. Patient assessment of bowel function during and after pelvic radiotherapy: results of a prospective phase III North Central Cancer Treatment Group clinical trial. J Clin Oncol. 2007 Apr 1;25(10):1255-9. doi: 10.1200/JCO.2006.09.0001. PMID 17401014
- [Result] Andreyev J. Gastrointestinal symptoms after pelvic radiotherapy: a new understanding to improve management of symptomatic patients. Lancet Oncol. 2007 Nov;8(11):1007-17. doi: 10.1016/S1470-2045(07)70341-8. PMID 17976611
- [Result] Kumagai T, Rahman F, Smith AM. The Microbiome and Radiation Induced-Bowel Injury: Evidence for Potential Mechanistic Role in Disease Pathogenesis. Nutrients. 2018 Oct 2;10(10):1405. doi: 10.3390/nu10101405. PMID 30279338
- [Result] Henson CC, Andreyev HJ, Symonds RP, Peel D, Swindell R, Davidson SE. Late-onset bowel dysfunction after pelvic radiotherapy: a national survey of current practice and opinions of clinical oncologists. Clin Oncol (R Coll Radiol). 2011 Oct;23(8):552-7. doi: 10.1016/j.clon.2011.04.002. Epub 2011 May 6. PMID 21550216
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Andreyev HJ, Vlavianos P, Blake P, Dearnaley D, Norman AR, Tait D. Gastrointestinal symptoms after pelvic radiotherapy: role for the gastroenterologist? Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1464-71. doi: 10.1016/j.ijrobp.2004.12.087. PMID 15927411
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338